CLINICAL TRIAL: NCT01499940
Title: Phase II Study to Assess Prevention of Oxaliplatin-induced Neurotoxicity Through the Vitamin D Pathway
Brief Title: Study to Assess Prevention of Oxaliplatin-induced Neurotoxicity Through Vitamin D Pathway
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Research cancelled - no funding identified.
Sponsor: Gerald Higa, PharmD. (Other)
Responsible Party: Sponsor-Investigator, Gerald Higa, PharmD., Associate Professor, West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WVU 11011
Record Dates: First submitted 2011-10-18; First posted 2011-12-26 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Neurotoxicity
Keywords: peripheral neuropathy; vitamin D status; oxaliplatin
MeSH Terms: conditions — Neurotoxicity Syndromes; Peripheral Nervous System Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D3 2000 IU/day (Experimental): Vitamin D3 2000 IU/day on day of 1st cycle of oxaliplatin; continue as long as patient treated with oxaliplatin and remains on study
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 will be administered at a dose of 2000 IU orally daily starting on day 1 of the first cycle of oxaliplatin. The vitamin will be continued at this dose and schedule for approximately 6 months if the patient is receiving oxaliplatin in the adjuvant setting and neither dosage nor interval has been modified for neurological toxicity. The duration of therapy if oxaliplatin is given for metastatic disease will vary. Nonetheless, the study vitamin will be continued using the same criteria as in the adjuvant setting.
  Other Names: Cholecalciferol

SUMMARY:
Many patients with cancer that are treated with a drug called oxaliplatin. This drug is used with other drugs to treat cancer. The drug can cause problems with the nerves in the hands and feet called peripheral neuropathy (a side effect of the drug). Peripheral neuropathy may make the hands and feet feel like they are tingling, have a burning feeling, and can cause pain. Almost all patients who receive oxaliplatin as part of their cancer treatment have peripheral neuropathy. Patients who do have this side effect usually have to take a lower dose of or stop taking the oxaliplatin even if the drug is helping their cancer.

So far there is not a lot of information about how to make this side effect better or help it go away completely. There is some information that low levels of Vitamin D in the blood might be linked to problems or diseases of the nervous system like multiple sclerosis or Parkinson's Disease. It is even thought that Vitamin D may help protect the cells in the nervous system. Because of this information, researchers want to see if giving patients Vitamin D while they are receiving the drug oxaliplatin to see if it helps prevent the side effect peripheral neuropathy.

Patients taking oxaliplatin who want to be in this study will take one Vitamin D capsule each day while they take oxaliplatin. Being in this study will not affect how the patient's cancer is treated. There are blood tests in the study to check Vitamin D levels and for a protein called nerve growth factor (NGF). The study team will carefully monitor the patients for any signs of oxaliplatin-related neurologic toxicity during the study.

DETAILED DESCRIPTION:
Oxaliplatin is used most frequently in patients with metastatic and early-stage colorectal cancers. It has been found that in the adjuvant setting, Oxaliplatin improves both disease free and overall survival. Despite these results, the use of Oxaliplatin is limited by the sensory neuropathy or numbness and tingling, that occurs in 80% -90% of patients. Some of these patients will develop irreversible and debilitating neuropathy, in which the drug may no longer be used to treat their cancer.

It is expected that this proposed study will provide new information for the role of Vitamin D in the pathogenesis of Oxaliplatin-induced neurotoxicity. The dynamic effects of Vitamin D on calcium and nerve growth factor plus the now recognized state of subclinical Vitamin D deficiency are compelling pieces of evidence that indicate this hormone may be in a pivotal position in the multifactorial pathogenesis of neurotoxic reactions induced by Oxaliplatin. The specific aim of the study is to determine the neuroprotective effects of Vitamin D.

Patients will receive Oxaliplatin at a dose of 80 mg/m2 at a physician determined frequency appropriate for the underlying malignancy, which can be any histological diagnosis of a malignant solid neoplasm involving the GI tract not restricted to the colon, rectum and esophagus. Blood will be collected to monitor the level of Vitamin D and nerve growth factor (NGF) at specific time points. Vitamin D levels will be checked once a month and NGF levels will be checked bi-weekly. These blood samples will be collected at the same time of the patients routine blood draws. Patients will take one capsule containing 2000 IUs of Vitamin D3 daily, beginning up to 7 days prior to the first dose of Oxaliplatin. Vitamin D3 will be provided to patients as long as they remain on the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologic diagnosis of a malignant solid neoplasm involving the gastrointestinal tract not necessarily restricted to the colon, rectum, and esophagus,
* Will receive oxaliplatin-based chemotherapy for the first time (previous treatment with non-oxaliplatin-based chemotherapy does not preclude eligibility),
* Have disease of any stage and will be treated according to established standards,
* Have a performance status (ECOG) of 2 or less,
* Have intact organ function as determined by laboratory tests of the kidney, liver, and bone marrow deemed appropriate to receive cytotoxic chemotherapy,
* Are 18 years of age or older, and
* Have signed a consent and information form to participate in the study.

Exclusion Criteria:

* Are pregnant (subjects of childbearing age will have a pregnancy test performed),
* Are taking calcitriol or have vitamin D levels that are >100 ng/dL,
* Are receiving medication for seizures, or
* Have pre-existing peripheral neuropathy grade >1.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Higa, PharmD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Kim JS, Ryu SY, Yun I, Kim WJ, Lee KS, Park JW, Kim YI. 1alpha,25-Dihydroxyvitamin D(3) Protects Dopaminergic Neurons in Rodent Models of Parkinson's Disease through Inhibition of Microglial Activation. J Clin Neurol. 2006 Dec;2(4):252-7. doi: 10.3988/jcn.2006.2.4.252. Epub 2006 Dec 20. PMID 20396528
- [Background] Wang JY, Wu JN, Cherng TL, Hoffer BJ, Chen HH, Borlongan CV, Wang Y. Vitamin D(3) attenuates 6-hydroxydopamine-induced neurotoxicity in rats. Brain Res. 2001 Jun 15;904(1):67-75. doi: 10.1016/s0006-8993(01)02450-7. PMID 11516412
- [Background] Bischoff-Ferrari HA, Giovannucci E, Willett WC, Dietrich T, Dawson-Hughes B. Estimation of optimal serum concentrations of 25-hydroxyvitamin D for multiple health outcomes. Am J Clin Nutr. 2006 Jul;84(1):18-28. doi: 10.1093/ajcn/84.1.18. PMID 16825677
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Heaney RP. Functional indices of vitamin D status and ramifications of vitamin D deficiency. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1706S-9S. doi: 10.1093/ajcn/80.6.1706S. PMID 15585791

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 2000 IU/Day
Started | 9
Completed | 0
Not Completed | 9
Not completed — Study was withdrawn before completion. | 9

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D3 2000 IU/Day
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Peripheral Neurotoxic Reactions
Description: NCI CTCAE Version 4.0
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 2000 IU/Day
Number analyzed (Participants) | 9
Participants | 5

ADVERSE EVENTS:
Arm/Group | Vitamin D3 2000 IU/Day
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes